CLINICAL TRIAL: NCT01395329
Title: Nebivolol and the Endothelin (ET)-1 System
Acronym: NETS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Christopher DeSouza, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: BYS-MD-57
Record Dates: First submitted 2011-06-09; First posted 2011-07-15 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Prehypertension; Hypertension
MeSH Terms: conditions — Prehypertension; Hypertension | interventions — Nebivolol; Metoprolol; cyclo(Trp-Asp-Pro-Val-Leu); BQ 788

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nebivolol (Active Comparator): Systolic and Diastolic blood pressure will be measured before and after randomization to12 weeks of Nebivolol. Forearm blood flow will be measured in response to 100 nmol/min of BQ-123, BQ-123+BQ788 (50 mol/min), Acetylcholine (4.0, 8.0, 16.0 ug/100 mL tissue/min), Sodium Nitroprusside (1.0, 2.0, 4.0 ug/100 mL tissue/min) and BQ-123+BQ-788+Acetylcholine (same doses as above) will be measured before and after the 12 weeks of nebivolol.
  Interventions: Drug: Nebivolol; Other: Forearm Blood Flow (FBF) response to BQ-123 (100 mol/min); Other: FBF response to BQ-123 (100 nmol/min)+BQ-788(50 nmol/min); Other: FBF response to Acetylcholine; Other: FBF response to Sodium Nitroprusside; Other: FBF response to BQ-123+BQ-788+ACh
- Metoprolol (Active Comparator): Systolic and Diastolic blood pressure will be measured before and after randomization to12 weeks of Metoprolol. Forearm blood flow will be measured in response to 100 nmol/min of BQ-123, BQ-123+BQ788 (50 mol/min), Acetylcholine (4.0, 8.0, 16.0 ug/100 mL tissue/min), Sodium Nitroprusside (1.0, 2.0, 4.0 ug/100 mL tissue/min) and BQ-123+BQ-788+Acetylcholine (same doses as above) will be measured before and after the 12 weeks of Metoprolol.
  Interventions: Drug: Metoprolol; Other: Forearm Blood Flow (FBF) response to BQ-123 (100 mol/min); Other: FBF response to BQ-123 (100 nmol/min)+BQ-788(50 nmol/min); Other: FBF response to Acetylcholine; Other: FBF response to Sodium Nitroprusside; Other: FBF response to BQ-123+BQ-788+ACh
- Placebo (Placebo Comparator): Systolic and Diastolic blood pressure will be measured before and after randomization to12 weeks of placebo. Forearm blood flow will be measured in response to 100 nmol/min of BQ-123, BQ-123+BQ788 (50 mol/min), Acetylcholine (4.0, 8.0, 16.0 ug/100 mL tissue/min), Sodium Nitroprusside (1.0, 2.0, 4.0 ug/100 mL tissue/min) and BQ-123+BQ-788+Acetylcholine (same doses as above) will be measured before and after the 12 weeks of placebo.
  Interventions: Drug: Placebo; Other: Forearm Blood Flow (FBF) response to BQ-123 (100 mol/min); Other: FBF response to BQ-123 (100 nmol/min)+BQ-788(50 nmol/min); Other: FBF response to Acetylcholine; Other: FBF response to Sodium Nitroprusside; Other: FBF response to BQ-123+BQ-788+ACh

INTERVENTIONS:
Drug: Nebivolol — 5 mg tablet to be taken by mouth once per day for 12 weeks
  Other Names: Bystolic
  Arms: Nebivolol
Drug: Metoprolol — 100 mg tablet to be taken by mouth once per day for 12 weeks
  Other Names: Toprol-XL
  Arms: Metoprolol
Drug: Placebo — gelatin capsule to be taken by mouth once per day for 12 weeks
  Arms: Placebo
Other: Forearm Blood Flow (FBF) response to BQ-123 (100 mol/min) — The forearm blood flow response to the endothelin (ET) -1 A receptor blocker BQ-123 (100 nmol/min) for 60 minutes at baseline and at 12 weeks.
  Other Names: BQ-123
Other: FBF response to BQ-123 (100 nmol/min)+BQ-788(50 nmol/min) — The FBF response to the nonselective endothelin (ET) -1 receptor blockade BQ-123 (100 nmol/min) + BQ-788 (50 nmol/min)for 60 minutes at baseline and at 12 weeks.
  Other Names: BQ-123+BQ-788
Other: FBF response to Acetylcholine — The FBF response to the endothelium-dependent vasodilator ACh (4, 8 and 16 ug/100 mL tissue/min) at baseline and at 12 weeks.
  Other Names: ACh
Other: FBF response to Sodium Nitroprusside — The FBF response to the endothelium independent vasodilator NTP (1,2 and 4 ug/100 mL tissue/min) at baseline and at 12 weeks.
  Other Names: NTP
Other: FBF response to BQ-123+BQ-788+ACh — The FBF response to the nonselective endothelin (ET) -1 receptor blockade BQ-123 (100 nmol/min) + BQ-788 (50 nmol/min)for 60 minutes at baseline and at 12 weeks.
  Other Names: BQ-123+BQ-788+ACh

SUMMARY:
The investigators hypothesize that nebivolol will reduce ET-1-mediated vasoconstrictor tone in adult humans with elevated blood pressure to a greater extent than either metoprolol or placebo.

DETAILED DESCRIPTION:
1. The investigators hypothesize that nebivolol will reduce ET-1-mediated vasoconstrictor tone in adult humans with elevated blood pressure to a greater extent than either metoprolol or placebo.
2. The investigators further hypothesize that reducing ET-1 vasoconstrictor activity contributes to the improvement in endothelial vasodilator function associated with nebivolol.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be men and women of all races and ethnic backgrounds aged 45-65 years.
* Subjects will be prehypertensive/hypertensive defined as resting systolic blood pressure >130 mmHg and < 160 mm Hg and/or diastolic blood pressure >80 mmHg and < 100 mm Hg.
* All of the women in the study will be postmenopausal (at least 1 year from last menstrual cycle) and not receiving hormone replacement therapy (HRT) currently or in the preceding 3-year period.
* Lastly, candidates will be sedentary as determined from the Stanford Physical Activity Questionnaire (<35 kcal/wk) and will not have engaged in any program of regular physical activity for at least 1 year prior to the study.

Exclusion Criteria:

* Candidates who smoke (currently or in the past 7 years), report more than low-risk alcohol consumption as defined as no more than 14 standard drinks/wk and no more than 4 standard drinks/day for men and 7 standard drinks/wk and 3 standard drinks/day for women (a standard drink is defined as 12 ounces of beer, 5 ounces of wine, 1½ ounces of 80-proof distilled spirits)
* Potential candidates who are taking cardiovascular-acting (i.e. statins, blood pressure medication an aspirin) medications will not be eligible.
* Fasting plasma glucose >126 mg/dL.
* Potential candidates with a resting heart rate of < 50 beats/minute will be excluded.
* Use of hormone replacement therapy.
* In hypertensive subjects, a seated systolic blood pressure greater than 160 mmHg or a seated diastolic blood pressure greater than 100 mmHg.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-05; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A DeSouza, Ph.D., Principal Investigator — University of Colorado at Boulder
Locations (1):
- UC-Boulder Clinical and Translational Research Center, Boulder, Colorado, United States

REFERENCES:
- [Derived] Diehl KJ, Stauffer BL, Dow CA, Bammert TD, Brunjes DL, Greiner JJ, DeSouza CA. Chronic Nebivolol Treatment Suppresses Endothelin-1-Mediated Vasoconstrictor Tone in Adults With Elevated Blood Pressure. Hypertension. 2016 Jun;67(6):1196-204. doi: 10.1161/HYPERTENSIONAHA.115.06979. Epub 2016 Apr 25. PMID 27113048

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nebivolol | Metoprolol | Placebo
Started | 14 | 14 | 14
Completed | 14 | 14 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Metoprolol | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 14 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 14 | 42
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (5.3) | 55 (4.1) | 56 (5.9) | 56 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 5 | 16
  Male | 8 | 9 | 9 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 14 | 14 | 42

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Time Frame: Systolic blood pressure was measured before the 12 week drug or placebo intervention and after the 12 week drug or placebo intervention.
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Before Nebivolol: Before randomization to Nebivolol
- After Nebivolol: Nebivolol: 5 mg tablet to be taken by mouth once per day for 12 weeks
- Before Metoprolol: Before randomization to Metoprolol
- After Metoprolol: Metoprolol: 100 mg tablet to be taken by mouth once per day for 12 weeks
- Before Placebo: Before randomization to placebo
- After Placebo: Placebo: gelatin capsule to be taken by mouth once per day for 12 weeks
Arm/Group | Before Nebivolol | After Nebivolol | Before Metoprolol | After Metoprolol | Before Placebo | After Placebo
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
mmHg | 144 (6.6) | 126 (7.8) | 140 (6.1) | 125 (9.3) | 139 (4.9) | 134 (8.3)

2. Primary Outcome: Diastolic Blood Pressure
Time Frame: Diastolic blood pressure was measured before the 12 week drug or placebo intervention and after the 12 week drug or placebo intervention.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Before Nebivolol | After Nebivolol | Before Metoprolol | After Metoprolol | Before Placebo | After Placebo
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
mmHg | 89 (5.2) | 77 (5.3) | 90 (7.6) | 77 (4.8) | 86 (7.7) | 83 (7.3)

3. Primary Outcome: Percent Change in Forearm Blood Flow (FBF) Response to BQ-123 (100 Nmol/Min)
Description: Forearm blood flow (FBF) was measured via strain-gauge venous occlusion plethysmography at rest and every 10 minutes thereafter for 60 minutes. The average percent change for before and after either drug or placebo was calculated as the FBF at (each time point-resting value)/resting value and multiplied by 100 to calculate the percent change. The baseline or resting value was measured before the start of each drug infusion.
Time Frame: Forearm blood flow was measured at 0-60 minutes before the 12 week drug or placebo intervention and 0-60 minutes after the 12 week drug or placebo intervention.
Measure: Mean (Standard Error); unit: percent change from baseline
Arm/Group | Before Nebivolol | After Nebivolol | Before Metoprolol | After Metoprolol | Before Placebo | After Placebo
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
percent change from baseline
  BQ-123 10 min | 10.2 (2.6) | -1.0 (1.7) | 10.0 (3.7) | 11.1 (2.8) | 13.1 (4.6) | 15.7 (3.0)
  BQ-123 20 min | 17.4 (3.3) | 6.0 (3.3) | 18.0 (4.7) | 18.7 (3.2) | 20.4 (3.1) | 14.7 (3.9)
  BQ-123 30 min | 22.3 (5.1) | -1.1 (3.3) | 23.0 (4.6) | 21.1 (4.8) | 26.8 (5.1) | 23.3 (4.5)
  BQ-123 40 min | 25.6 (6.3) | 3.8 (3.2) | 28.4 (4.9) | 28.9 (3.8) | 23.9 (4.3) | 25.7 (3.9)
  BQ-123 50 min | 25.8 (4.6) | 6.1 (3.6) | 31.4 (5.9) | 27.7 (4.8) | 29.0 (5.6) | 26.5 (4.5)
  BQ-123 60 min | 27.0 (6.4) | 1.1 (4.5) | 34.4 (5.7) | 30.6 (5.5) | 33.8 (5.3) | 30.4 (3.7)

4. Primary Outcome: Percent Change in FBF Response to BQ-123 (100 Nmol/Min) + BQ-788 (50 Nmol/Min)
Description: as for outcome 3
Time Frame: Forearm blood flow was measured 0-120 minutes before the 12 week drug or placebo intervention and 0-120 minutes after the 12 week drug or placebo intervention.
Measure: Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Before Nebivolol | After Nebivolol | Before Metoprolol | After Metoprolol | Before Placebo | After Placebo
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
Percent change from baseline
  BQ-123 10 min | 10.2 (2.6) | -1.0 (1.7) | 10.0 (3.7) | 11.1 (2.8) | 13.1 (4.6) | 15.7 (3.0)
  BQ-123 20 min | 17.4 (3.3) | 6.0 (3.3) | 18.0 (4.7) | 18.7 (3.2) | 20.4 (3.1) | 14.7 (3.9)
  BQ-123 30 min | 22.3 (5.1) | -1.1 (3.3) | 23.0 (4.6) | 21.1 (4.8) | 26.8 (5.1) | 23.3 (4.5)
  BQ-123 40 min | 25.6 (6.3) | 3.8 (3.2) | 28.4 (4.9) | 28.9 (3.8) | 23.9 (4.3) | 25.7 (3.9)
  BQ-123 50 min | 25.8 (4.6) | 6.1 (3.6) | 31.4 (5.9) | 27.7 (4.8) | 29.0 (5.6) | 26.5 (4.5)
  BQ-123 60 min | 27.0 (6.4) | 1.1 (4.5) | 34.4 (5.7) | 30.6 (5.5) | 33.8 (5.3) | 30.4 (3.7)
  BQ-123+BQ-788 70 min | 44.0 (6.9) | 9.2 (3.7) | 33.2 (6.9) | 37.8 (5.7) | 37.5 (8.3) | 38.0 (7.5)
  BQ-123+BQ-788 80 min | 41.3 (7.0) | 16.1 (8.2) | 44.7 (7.3) | 32.2 (7.3) | 42.6 (9.5) | 45.0 (7.9)
  BQ-123+BQ-788 90 min | 39.5 (7.1) | 21.8 (9.2) | 49.8 (9.5) | 47.4 (6.9) | 46.4 (8.9) | 47.1 (7.4)
  BQ-123+BQ-788 100 min | 47.4 (7.8) | 22.3 (8.5) | 47.5 (7.4) | 42.0 (7.6) | 57.1 (9.5) | 53.4 (8.5)
  BQ-123+BQ-788 110 min | 47.6 (8.5) | 18.9 (7.0) | 57.8 (10.4) | 48.1 (7.6) | 57.8 (7.8) | 52.8 (9.3)
  BQ-123+BQ-788 120 min | 57.6 (9.0) | 20.4 (7.6) | 64.6 (9.8) | 55.4 (7.1) | 57.9 (9.5) | 49.5 (10.3)

5. Primary Outcome: FBF Response to Acetylcholine (ACh)
Description: FBF was measured via strain-gauge occlusion plethysmography at rest and in response to ACh (4.0, 8.0 and 16.0 ug/100 mL tissue/min) for 5 minutes at each dose. Flows during the last minute of rest and each drug dose were measured and the mean value reported.
Time Frame: Forearm blood flow was measured before the 12 week drug or placebo intervention and after the 12 week drug or placebo intervention.
Measure: Mean (Standard Error); unit: mL/100 mL tissue/min
Arm/Group | Before Nebivolol | After Nebivolol | Before Metoprolol | After Metoprolol | Before Placebo | After Placebo
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
mL/100 mL tissue/min
  Baseline | 5.2 (0.3) | 4.9 (0.4) | 5.3 (0.5) | 5.6 (0.5) | 4.8 (0.2) | 5.1 (0.3)
  ACh 4.0 | 12.1 (0.8) | 13.9 (0.9) | 12.4 (1.0) | 12.0 (1.0) | 11.4 (0.6) | 13.2 (0.7)
  ACh 8.0 | 12.7 (0.8) | 15.0 (0.8) | 13.1 (1.1) | 13.2 (1.1) | 12.0 (0.6) | 13.7 (0.6)
  ACh 16.0 | 13.3 (0.8) | 16.4 (0.6) | 13.8 (1.1) | 14.1 (1.1) | 12.7 (0.8) | 13.9 (0.7)

6. Primary Outcome: FBF Response to Sodium Nitroprusside
Description: FBF was measured via strain-gauge occlusion plethysmography at rest and in response to sodium nitroprusside (1.0, 2.0 and 4.0 ug/100 mL tissue/min) for 5 minutes at each dose. Flows during the last minute of rest and each drug dose were measured and the mean value reported.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: mL/100 mL tissue/min
Arm/Group | Before Nebivolol | After Nebivolol | Before Metoprolol | After Metoprolol | Before Placebo | After Placebo
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
mL/100 mL tissue/min
  Baseline | 5.2 (0.4) | 4.7 (0.3) | 4.9 (0.3) | 5.7 (0.5) | 5.2 (0.3) | 5.2 (0.3)
  Sodium Nitroprusside 1.0 | 13.5 (1.2) | 13.7 (1.0) | 14.1 (1.3) | 14.3 (1.2) | 12.8 (0.7) | 13.7 (0.8)
  Sodium Nitroprusside 2.0 | 15.3 (1.3) | 15.2 (1.0) | 14.9 (1.3) | 15.1 (1.1) | 14.4 (0.8) | 15.3 (0.8)
  Sodium Nitroprusside 4.0 | 15.9 (1.2) | 16.4 (1.1) | 15.8 (1.3) | 16.0 (1.0) | 15.8 (0.8) | 16.1 (0.9)

7. Primary Outcome: FBF Response to ACh in the Absence or Presence of Nonselective Endothelin A/B Blockade (BQ-123+BQ-788)
Description: FBF was measured via strain-gauge occlusion plethysmography at rest and in response to BQ-123+BQ-788 +ACh (4.0, 8.0 and 16.0 ug/100 mL tissue/min) for 5 minutes at each dose. Flows during the last minute of rest and each drug dose were measured and the mean value reported.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: mL/100 mL tissue/min
Arm/Group | Before Nebivolol | After Nebivolol | Before Metoprolol | After Metoprolol | Before Placebo | After Placebo
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
mL/100 mL tissue/min
  Baseline | 5.0 (0.3) | 4.7 (0.3) | 5.5 (0.4) | 6.0 (0.5) | 4.9 (0.2) | 5.1 (0.3)
  ACh 4.0 | 11.7 (0.8) | 13.8 (0.9) | 13.1 (1.1) | 12.4 (1.1) | 11.7 (0.6) | 13.3 (0.7)
  ACh 8.0 | 12.3 (0.7) | 15.0 (0.7) | 13.7 (1.2) | 13.7 (1.2) | 12.3 (0.7) | 13.7 (0.7)
  ACh 16.0 | 12.9 (0.7) | 16.1 (0.5) | 14.5 (1.2) | 14.7 (1.2) | 13.0 (0.8) | 13.9 (0.8)
  Baseline+BQ123/788 | 6.4 (0.5) | 5.8 (0.7) | 6.7 (0.4) | 7.4 (0.7) | 6.1 (0.4) | 5.6 (0.4)
  ACh 4.0+BQ-123/788 | 14.6 (0.7) | 13.7 (0.9) | 16.1 (1.3) | 16.5 (1.3) | 13.5 (1.0) | 15.3 (0.9)
  ACh 8.0+BQ-123/788 | 15.3 (0.7) | 14.5 (0.8) | 17.1 (1.2) | 17.6 (1.2) | 15.1 (0.9) | 16.5 (0.9)
  ACh 16.0+BQ-123/788 | 15.9 (0.6) | 15.0 (0.7) | 17.9 (1.3) | 18.2 (1.2) | 16.2 (0.9) | 17.3 (1.0)

ADVERSE EVENTS:
Arm/Group | Nebivolol | Metoprolol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No